CLINICAL TRIAL: NCT01742767
Title: Randomized Phase II Trial of Three-weekly Cisplatinum and Pemetrexed Versus Split-dose d1 and d8 Cisplatinum and Pemetrexed In Advanced and Inoperable Non-squamous Non-small-cell Lung Cancer (NSCLC)
Brief Title: Cisplatinum/Pemetrexed Versus Split-dose Cisplatinum/Pemetrexed In NSCLC
Acronym: PemSplitCisp
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Mathias Hoiczyk, Physician, Universität Duisburg-Essen
Model: Parallel | Purpose: Treatment
Other Study IDs: 2011-001963-37
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: NSCLC
Keywords: NSCLC; split dose Cisplatinum; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cis (D1) + Pem (D1) (Active Comparator): Cisplatinum 75 mg/m2 d 1 Pemetrexed 500 mg/m2 d 1 q d 21
  Interventions: Drug: Cisplatinum; Drug: Pemetrexed
- CIS (D1+8) + Pem (D!) (Experimental): Cisplatinum 40 mg/m2 d 1 + d 8 Pemetrexed 500 mg/m2 d 1 q d 21
  Interventions: Drug: Cisplatinum; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cisplatinum
Drug: Pemetrexed

SUMMARY:
Cisplatinum and pemetrexed (ALIMTA®) has become an effective first-line regimen for advanced and inoperable non-squamous NSCLC without somatic activating mutations of epidermal growth factor receptor (EGFR). In the standard regimen the cisplatinum dose is 75 mg/m2 on day 1 of a 21-day cycle. Due to the high platinum-dose patients do need a strict hyperhydration and often have to be hospitalized for survey. Split-dose cisplatinum with two administrations on Day 1 and 8 of a 21-day-cycle has already been administered in other platin-containing chemotherapy regimens (cis/gem cis/nav cis/paclitaxel cis/docetaxel) with favourable toxicity profiles and generally with an excellent patient compliance.

DETAILED DESCRIPTION:
There is a current need to develop a split-dose cisplatinum regimen in combination with pemetrexed with high efficacy, excellent treatment compliance, administration convenience and the possibility to open up easier outpatient administration of the chemotherapy protocol. Dosing of cisplatinum at 40 mg/m2 d 1 and day 8 seems to be very effective and useful for this strategy. The current trial will address this issue within a prospective randomized phase-II trial. Treatment will be given on day 1 and 8 in the split-dose arm. A comparator arm of the current three-weekly higher cisplatinum schedule will be added to this study. For evaluation of this strategy observation of the toxicity/efficacy ratio within this trial will be of major importance. Efficacy will be analyzed by objective response rate, symptom control and life-quality. Toxicity will be looked at with treatment toxicity, treatment compliance and adherence to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be included in the study only if they meet all of the following criteria:

  1. Histologically or cytologically confirmed diagnosis of non-squamous-cell non-small cell lung cancer (NSCLC) Stage IV (American Joint Committee on Cancer Staging Criteria [AJCC], Version 7, 2009)
  2. No prior systemic chemotherapy for lung cancer
  3. At least one unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST; version 1.1, Eisenhauer et al. 2009), longest diameter ≥10 mm with computed tomography (CT) scan [CT scan slice thickness no greater than 5 mm] , or ≥ 20 mm with chest x-ray. Positron emission tomography (PET) scans and ultrasounds should not be used.
  4. ECOG performance status of 0 or 1 (Oken et al. 1982)
  5. ≥ 18 years of age < 75 years
  6. Adequate organ function,
  7. Prior radiation therapy allowed to <25% of the bone marrow (Cristy and Eckerman 1987). Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.
  8. Patient must understand and sign an informed consent document before the start of specific protocol procedures.
  9. A pretreatment FFPE tumour biopsy must be available for central biomarker analysis. If consented by the patient and clinically feasible, a fresh pretreatment biopsy is obtained and submitted for central biomarker analysis.
  10. Female patients with childbearing potential must use highly effective methods of contraception (combined oral contraceptives, hormon-releasing intrauterine contraceptive device, hormonal contraceptive implants, hormonal contraceptive injectables) or have sexual intercourse with a vasectomised partner only during and for 6 months after the study and their pregnancy test must be negative within 7 days prior to study enrollment.

      A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 year or unless she is surgically sterile.

      Male patients must agree to use condoms during the study and for 6 months after the study if their partner is of childbearing potential and does not use highly effective method of contraception.
  11. Estimated life expectancy of 12 weeks
  12. Patient compliance and geographic proximity that allow adequate follow up.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  1. Active participation in other clinical studies or treatment with any experimental drug within 30 days prior to study enrollment or during study participation.
  2. Patients with known somatic activating mutations of EGFR, as these patients should be offered EGFR- tyrosine kinase inhibitor (EGFR-TKI) treatment as first-line therapy. Detection of EGFR mutations and additional somatic mutations with relation to treatment will be performed centrally at the Universitätsklinikum Essen. In case immediate treatment initiation is required for medical reasons (such as superior vena cava syndrome, severely symptomatic disease) patients may be enrolled before results from EGFR testing are available. As EGFR-TKI treatment is equally effective in second-line therapy, such patients may remain on study treatment if a clinical benefit is derived.
  3. Peripheral neuropathy of ³CTCAE Grade 1
  4. Inability to comply with protocol or study procedures
  5. A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
  6. A serious cardiac condition, such as myocardial infarction within 6 months prior to study enrollment, symptomatic coronary artery disease, cardiac arrhythmia, or other heart disease, as defined by the New York Heart Association Class III or IV (functional capacity)
  7. Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
  8. Documented brain metastases unless the patient has completed successful local therapy for central nervous system metastases and has been off of corticosteroids for at least 4 weeks before enrollment. Brain imaging is required in symptomatic patients to rule out brain metastases,but is not required in asymptomatic patients
  9. The effect of third space fluid, such as pleural effusion and ascites, on pemetrexed is unknown. In patients with clinically significant third space fluid, consideration should be given to draining the effusion prior to pemetrexed administration.
  10. Significant weight loss (that is 10%) over the previous 6 weeks before study entry
  11. Significant hearing function impairment, especially high-frequency hearing function impairment
  12. Any active or uncontrolled infection
  13. Concurrent administration of any other antitumour therapy
  14. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose <1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
  15. Inability or unwillingness to take folic acid or vitamin B12 supplementation
  16. Inability to take corticosteroids
  17. Hypersensitivity to cisplatinum or to any other platinum compound
  18. Hypersensitivity to pemetrexed or to any of the excipients of ALIMTA®
  19. Pregnant or breast-feeding patient
  20. Yellow fever vaccination within the 30 days previous to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-11; Primary Completion 2014-05 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Eberhardt, MD, Principal Investigator — Universital hospital essen
Locations (1):
- University hospital essen, Essen, North Rhine-Westphalia, Germany